CLINICAL TRIAL: NCT06098963
Title: Preliminary Outcomes of Sacral Neuromodulation Applications; Tertiary-Center Experience in Turkey
Status: Completed | Type: Observational
Sponsor: Cigli Regional Training Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Ozan Horsanalı, Associated professor, Cigli Regional Training Hospital
Other Study IDs: CigliRTH
Record Dates: First submitted 2023-10-15; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Sacral Neuromodulation
Keywords: Sacral neuromodulation; Overactive bladder; Urinary incontinence; Fecal incontinence; Lower urinary tract dysfunction
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: sacral neuromodulation — sacra neuromodulator implantation outcomes

SUMMARY:
to report our patients' outcomes of SNM in tertiary health centres in Turkey

DETAILED DESCRIPTION:
We retrospectively analyzed 18 patients who underwent SNM for urinary or bowel dysfunction between 2017 and 2022 in our clinic. We excluded 2 patients due to non-effective responses after the test period. After local ethics committee approval was obtained from our institute (Number and date: 21-12.1T/14). Patient characteristics and demographic data including age, gender, indications to the SNM, age at diagnosis, and comorbidities were collected from our Hospital patients' record system. Urinary functions were evaluated by the ICIQ-SF questionnaire form. Patients' diagnosis, implantation duration, complications, and improvement of symptoms were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with urinary incontinence
* Patients diagnosed with faecal incontinence
* Patients diagnosed with interstitial cystitis

Exclusion Criteria:

* Presence of urinary infection
* Presence of previous incontinence surgery
* Presence of 2nd motor neurone disease
* Inability of detrusor muscle contraction activity
* Previous radical cystoprostatectomy history
* Presence of bladder outlet obstruction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with urinary or faecal incontinence and interstitial cystitis who are unresponsible for medical therapy between the age of 18-85.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Recovery of urinary or fecal incontinence | 1 year
  Significant decrease in urinary or fecal incontinence episode

SECONDARY OUTCOMES:
increase in the score of ICIQ-SF questionnaire | 1 year
  improvement of quality of life and increase in the score of ICIQ-SF questionnaire

IPD SHARING:
Plan to Share IPD: No